CLINICAL TRIAL: NCT01611519
Title: Optimal Timing of Foley Catheter Removal in Patients Undergoing Thoracic Surgery With Epidural Analgesia: A Randomized, Controlled Trial
Brief Title: Early or Late Foley Removal After Thoracotomy
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark Allen, MD, Mayo Clinic
Other Study IDs: 11-006618
Record Dates: First submitted 2012-06-01; First posted 2012-06-05 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Urinary Tract Infections
Keywords: urinary bladder; urinary catheterization; epidural analgesia; catheters, indwelling
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Early (within 48 hours of surgery): Patients will have their urinary catheter removed within 48 hours of surgery
- Late (6 hours after epidural removal): Patients will have their urinary catheter removed 6 hours after their epidural is removed

SUMMARY:
Is the early removal of Foley catheter safe in patients undergoing general thoracic surgery with an epidural catheter in place?

DETAILED DESCRIPTION:
We hypothesis that removing the foley catheter within 48 hours after a thoracotomy in patients that have an epidural catheter will result in an increase in the rate of urinary infections and the need for reinsertion of the foley. We have designed a randomized trial to test this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* epidural catheter after thoracic surgery
* foley in place

Exclusion Criteria:

* < 18 years of age
* death in hospital within 30 days of the operation
* length of hospital stay is less than 48 hours
* epidural catheter is removed before the 3rd postoperative day
* patients who have a suprapubic catheter or no bladder
* patients who require a urologist or a urologic technician to insert the Foley catheter at the time of surgery
* patients who were being intermittently catheterized before surgery
* patients with a known urinary tract infection preoperatively
* patients required to keep Foley in since they required close monitoring of urinary output

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing thoracic surgery at the Mayo Clinic
Sampling Method: Probability Sample
Enrollment: 375 (Actual)
Dates: Start 2011-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Need for insertion of catheter after Foley removed. | participants will be followed for the duration of hospital stay, an expected average of 5 weeks

SECONDARY OUTCOMES:
Development of urinary tract infection | participants will be followed for the duration of hospital stay, an expected average of 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Allen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ellahi A, Stewart F, Kidd EA, Griffiths R, Fernandez R, Omar MI. Strategies for the removal of short-term indwelling urethral catheters in adults. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD004011. doi: 10.1002/14651858.CD004011.pub4. PMID 34184246